CLINICAL TRIAL: NCT02127567
Title: The Evaluation of a CONSORT Based Online Writing Tool: a Randomized Controlled Trial
Brief Title: The Evaluation of a CONSORT Based Online Writing Tool
Acronym: COBWEB
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Other
Other Study IDs: RAV009
Record Dates: First submitted 2014-04-29; First posted 2014-04-30 (Estimated); Results first posted 2015-03-20 (Estimated); Last update posted 2023-11-21 (Actual); Status verified 2014-04

CONDITIONS: Focus of Study = Medical Writing
Keywords: medical writing, reporting, randomized controlled trial

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Online writing tool (Experimental): Participants will be provided the corresponding CONSORT item(s), key elements from the explanation and elaboration of the CONSORT 2010 and NPT extension along with examples of good reporting
  Interventions: Other: online writing tool
- writing with no specific support. (Other): The control intervention will only consist of the title of the domain and a large text box where the participant will be asked to describe this part of the study for their study protocol. The participant will also have the option to indicate any important or necessary information that is not available in the provided study protocol.
  Interventions: Other: writing with no specific support

INTERVENTIONS:
Other: online writing tool — The writing tool contained the main CONSORT item and extension items for non pharmacological treatments along with bullet points indicating key elements to report from the explanation and elaboration publications of the CONSORT. Participants were also instructed to detail information they felt important to report but that was not available in the study protocol they were provided.
  Arms: Online writing tool
Other: writing with no specific support — The control tool simply provided the domain or section heading with a space too write. Similar to for the experimental intervention, participants were to indicate information they felt important to report but unavailable in the provided study protocols.
  Arms: writing with no specific support.

SUMMARY:
Introduction: Inadequate reporting is a frequent cause of waste of research. For example, essential information for evaluating the risk of bias such as the method of randomization is lacking in 75% of published randomized controlled trials (RCTs), and over 30% of reports do not provide sufficient details to allow replication of the treatment evaluated in the trial in clinical practice. To overcome this issue, the CONSORT statement, an evidence-based, minimum set of recommendations for reporting RCTs was developed in 1996. These guidelines have since been updated in 2001 and more recently in 2010. In addition, extensions to the main CONSORT statement have been developed to give additional guidance for RCTs with specific designs (eg cluster), data (eg harm), and interventions (eg nonpharmacologic treatments). Many journals endorse the CONSORT statement. Some journals provide recommendations to authors to follow the CONSORT guidelines and some editors enforce the use of the CONSORT guidelines by requesting authors to submit a checklist in either the submission or acceptance stage. Nevertheless, inadequate reporting remains.

Our objective is to evaluate the impact of the CONSORT based online writing tool on the completeness of reporting.

DETAILED DESCRIPTION:
Context Inadequate reporting is a frequent cause of waste of research. For example, essential information for evaluating the risk of bias such as the method of randomization is lacking in 75% of published randomized controlled trials (RCTs), and over 30% of reports do not provide sufficient details to allow replication of the treatment evaluated in the trial in clinical practice. To overcome this issue, the CONSORT statement, an evidence-based, minimum set of recommendations for reporting RCTs was developed in 1996. These guidelines have since been updated in 2001 and more recently in 2010. In addition, extensions to the main CONSORT statement have been developed to give additional guidance for RCTs with specific designs (eg cluster), data (eg harm), and interventions (eg nonpharmacologic treatments). Many journals endorse the CONSORT statement. Some journals provide recommendations to authors to follow the CONSORT guidelines and some editors enforce the use of the CONSORT guidelines by requesting authors to submit a checklist in either the submission or acceptance stage. Nevertheless, inadequate reporting remains.

Hypothesis We hypothesize that to improve reporting, the CONSORT guidelines must be implemented at the stage of the writing of the manuscript instead of at the stage of journal submission or peer review process. We developed a CONSORT based online writing tool to improve the completeness of reporting. This tool focuses on some domains of the methods section of a 2-arm parallel group randomized controlled trial evaluating pharmacologic or nonpharmacologic treatment.

Objective Our objective is to evaluate the impact of the CONSORT based online writing tool on the completeness of reporting.

Methods Study design: We will perform a "split-manuscript" randomized controlled trial, adapted from the split-body design. We will consider 6 domains of the methods section: trial design, randomization, blinding, participants, interventions, and outcomes. The unit of randomization will be the domain and the allocation ratio 1:1. Each study participant will receive the experimental intervention (the tool) for 3 of the 6 domains and the control intervention (no tool) for thther 3 domains.

Participants: Masters and doctoral students Intervention: The use of the online writing tool for writing the methods section of an article from an RCT protocol.

Comparator: The writing the methods section of an article from an RCT protocol with no specific support.

Primary outcome: The primary outcome will be the average score for completeness of reporting.

Number of participants expected: 40

ELIGIBILITY:
Inclusion Criteria

* Adults
* Masters or doctoral students

Exclusion criteria

* not in the field of medical research
* not adults
* no masters or doctoral level education

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2014-04; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Isabelle Boutron, Professor, Study Director — Public hospitals of Paris (APHP)
Locations (1):
- Hotel Dieu, 1, place du parvis de notre dame, Paris, France

REFERENCES:
- [Derived] Barnes C, Boutron I, Giraudeau B, Porcher R, Altman DG, Ravaud P. Impact of an online writing aid tool for writing a randomized trial report: the COBWEB (Consort-based WEB tool) randomized controlled trial. BMC Med. 2015 Sep 15;13:221. doi: 10.1186/s12916-015-0460-y. PMID 26370288

RESULTS

PARTICIPANT FLOW:
Groups:
- All Participants: All participants were asked to write the six parts or 'domains' of the methods section describing a randomized controlled trial. Each participant completed 3 parts or 'domains' with the tool and 3 without.
  online writing tool: The writing tool contained the main CONSORT item and extension items for non pharmacological treatments along with bullet points indicating key elements to report from the explanation and elaboration publications of the CONSORT. Participants were also instructed to detail information they felt important to report but that was not available in the study protocol they were provided.
Period: Overall Study
Arm/Group | All Participants
Started | 41 (41 participants completed 246 domains, 3 domains were completed with the tool per participant)
Completed | 41
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Forty-one masters and doctoral students participated. Participants median age was 29 with an interquartile range of 26 to 33. Just slightly over the majority were female, 24 (58.5%). And just slightly over the majorirty were already familiar with reporting guidelines, 24 (58.5%).
Arm/Group | All Participants
Number analyzed (Participants) | 41
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 29 [26 to 33]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24
  Male | 17
Education [Number; unit: participants] — doctoral vs masters students
  participants
    doctoral students | 14
    masters students | 27
Familiar with guidelines [Number; unit: participant]
  Familiar with guidelines | 24
  Not familiar with guidelines | 17
Frequency reading RCTs [Count of Participants; unit: Participants]
  More than once a year | 30
  once a month | 6
  Once a week | 5
Experience writing RCTs [Count of Participants; unit: Participants] | 7
Taught about RCTs [Count of Participants; unit: Participants] | 38
Previously involved in RCTs [Count of Participants; unit: Participants] | 18
Comfortable with English [Count of Participants; unit: Participants] | 26

OUTCOME MEASURES:

1. Primary Outcome: The Primary Outcome Will be the Average Score for Completeness of Reporting on a Scale of 0-10.
Description: Completeness of reporting will be determined according to a grading rubric individualized to each study protocol, 0 being the lowest and 10 the highest
Time Frame: one time measure after a four-hour writing session
Measure: Mean (Standard Deviation); unit: units on a scale
Units Other Than Participants: domains
Groups:
- Online Writing Tool, Experimental Arm: Participants will be provided the corresponding CONSORT item(s), key elements from the explanation and elaboration of the CONSORT 2010 and NPT extension along with examples of good reporting
  online writing tool: The writing tool contained the main CONSORT item and extension items for non pharmacological treatments along with bullet points indicating key elements to report from the explanation and elaboration publications of the CONSORT. Participants were also instructed to detail information they felt important to report but that was not available in the study protocol they were provided.
- Writing With no Specific Support, Control Arm: The control intervention will only consist of the title of the domain and a large text box where the participant will be asked to describe this part of the study for their study protocol. The participant will also have the option to indicate any important or necessary information that is not available in the provided study protocol.
  writing with no specific support: The control tool simply provided the domain or section heading with a space too write. Similar to for the experimental intervention, participants were to indicate information they felt important to report but unavailable in the provided study protocols.
Arm/Group | Online Writing Tool, Experimental Arm | Writing With no Specific Support, Control Arm
Number analyzed (Participants) | 41 | 41
Number analyzed (domains) | 123 | 123
units on a scale | 7.1 (1.2) | 5.0 (1.6)
Statistical Analysis 1: Comparison: Online Writing Tool, Experimental Arm vs Writing With no Specific Support, Control Arm; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis; Mean Difference (Final Values) = 2.1, 95% CI 2-sided [1.5 to 2.7]

2. Secondary Outcome: The Score for Completeness of Reporting for Randomization
Description: The score for completeness of reporting (0-10) for the manuscript section randomization, 0 being the lowest and 10 the highest
Time Frame: one time measure after a four-hour writing session
Measure: Mean (Standard Deviation); unit: units on a scale
Units Other Than Participants: domains
Arm/Group | Online Writing Tool | Writing With no Specific Support.
Number analyzed (Participants) | 20 | 21
Number analyzed (domains) | 20 | 21
units on a scale | 8.4 (2.4) | 4.6 (2.9)
Statistical Analysis 1: Comparison: Online Writing Tool vs Writing With no Specific Support; Test type: Superiority or Other; p < 0.01, Mixed Models Analysis; Mean Difference (Final Values) = 3.8, 95% CI 2-sided [1.1 to 4.4]

3. Secondary Outcome: The Score for Completeness of Reporting for Blinding
Description: on a scale from 0 to 10, 0 being the lowest and 10 the highest
Time Frame: one time measure after a four-hour writing session
Measure: Mean (Standard Deviation); unit: units on a scale
Units Other Than Participants: domains
Arm/Group | Online Writing Tool, Experimental Arm | Writing With no Specific Support, Control Arm
Number analyzed (Participants) | 21 | 20
Number analyzed (domains) | 21 | 20
units on a scale | 6.9 (2.4) | 6.2 (2.3)
Statistical Analysis 1: Comparison: Online Writing Tool, Experimental Arm vs Writing With no Specific Support, Control Arm; Test type: Superiority or Other; p = 0.44, Mixed Models Analysis; Mean Difference (Final Values) = 0.7, 95% CI 2-sided [-0.7 to 2.0]

4. Secondary Outcome: The Score for Completeness of Reporting for Participants
Description: on a scale from 0 to 10, 0 being the lowest and 10 the highest
Time Frame: one time measure after a four-hour writing session
Measure: Mean (Standard Deviation); unit: units on a scale
Units Other Than Participants: domains
Arm/Group | Online Writing Tool, Experimental Arm | Writing With no Specific Support, Control Arm
Number analyzed (Participants) | 21 | 20
Number analyzed (domains) | 21 | 20
units on a scale | 6.7 (2.0) | 4.5 (2.4)
Statistical Analysis 1: Comparison: Online Writing Tool, Experimental Arm vs Writing With no Specific Support, Control Arm; Test type: Superiority or Other; p < 0.01, Mixed Models Analysis; Mean Difference (Final Values) = 2.2, 95% CI 2-sided [0.8 to 3.6]

5. Secondary Outcome: The Score for Completeness of Reporting for Interventions
Description: on a scale from 0 to 10, 0 being the lowest and 10 the highest
Time Frame: one time measure after a four-hour writing session
Measure: Mean (Standard Deviation); unit: units on a scale
Units Other Than Participants: domain
Arm/Group | Online Writing Tool, Experimental Arm | Writing With no Specific Support, Control Arm
Number analyzed (Participants) | 20 | 21
Number analyzed (domain) | 20 | 21
units on a scale | 7.1 (1.5) | 5.3 (2.0)
Statistical Analysis 1: Comparison: Online Writing Tool, Experimental Arm vs Writing With no Specific Support, Control Arm; Test type: Superiority or Other; p < 0.01, Mixed Models Analysis; Median Difference (Final Values) = 1.8, 95% CI 2-sided [0.7 to 2.9]

6. Secondary Outcome: The Score for Completeness of Reporting for Outcomes
Description: on a scale from 0 to 10, 0 being the lowest and 10 the highest
Time Frame: one time measure after a four-hour writing session
Measure: Mean (Standard Deviation); unit: units on a scale
Units Other Than Participants: domain
Arm/Group | Online Writing Tool, Experimental Arm | Writing With no Specific Support, Control Arm
Number analyzed (Participants) | 20 | 21
Number analyzed (domain) | 20 | 21
units on a scale | 6.1 (2.1) | 6.4 (3.0)
Statistical Analysis 1: Comparison: Online Writing Tool, Experimental Arm vs Writing With no Specific Support, Control Arm; Test type: Superiority; p = 0.78, Mixed Models Analysis; Mean Difference (Final Values) = -0.3, 95% CI 2-sided [-2.0 to 1.3]

7. Secondary Outcome: The Score for Completeness of Reporting for Trial Design
Description: on a scale from 0 to 10, 0 being the lowest and 10 the highest
Time Frame: one time measure after a four-hour writing session
Measure: Mean (Standard Deviation); unit: units on a scale
Units Other Than Participants: domain
Arm/Group | Online Writing Tool, Experimental Arm | Writing With no Specific Support, Control Arm
Number analyzed (Participants) | 21 | 20
Number analyzed (domain) | 21 | 20
units on a scale | 8.1 (2.3) | 2.7 (1.9)
Statistical Analysis 1: Comparison: Online Writing Tool, Experimental Arm vs Writing With no Specific Support, Control Arm; Test type: Superiority or Other; p < 0.01, Mixed Models Analysis; Mean Difference (Final Values) = 5.4, 95% CI 2-sided [4.1 to 6.7]

8. Secondary Outcome: Average Score for Completeness of Reporting of Essential Elements
Description: Completeness of reporting scores calculated based on essential elements to report, on a scale from 0 to 10, 0 being the lowest and10 the highest
Time Frame: one time four hour writing session
Measure: Mean (Standard Deviation); unit: units on a scale
Units Other Than Participants: domains
Arm/Group | Online Writing Tool, Experimental Arm | Writing With no Specific Support, Control Arm
Number analyzed (Participants) | 41 | 41
Number analyzed (domains) | 123 | 123
units on a scale | 7.8 (1.6) | 6.4 (2.3)
Statistical Analysis 1: Comparison: Online Writing Tool, Experimental Arm vs Writing With no Specific Support, Control Arm; Test type: Superiority or Other; p = 0.002, Mixed Models Analysis; Mean Difference (Final Values) = 1.4, 95% CI 2-sided [0.5 to 2.3]

ADVERSE EVENTS:
Arm/Group | Online Writing Tool, Experimental Arm | Writing With no Specific Support, Control Arm
Serious Adverse Events (participants affected / at risk) | 0/41 | 0/41
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

LIMITATIONS AND CAVEATS:
We considered only six domains of the methods section of a manuscript We lack a validated outcome measure to appropriately evaluate the quality of reporting in various contexts.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes